CLINICAL TRIAL: NCT01298622
Title: The Study of Structural and Functional Brain Abnormalities and the Association With the Genetic Polymorphism in the Core Family of OCD Patient
Brief Title: The Imaging Genetic Study of the Core Family of Obsessive-compulsive Disorder (OCD) Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kunming Medical University (Other)
Responsible Party: Principal Investigator, Yuqi Cheng, prof., Kunming Medical University
Other Study IDs: OCD001
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: OCD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — perapheral blood DNA of all participants
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- controls
- OCD patients
- OCD parents

SUMMARY:
To investigate the structural/functional abnormalities and the possible genetic endophenotypes of Obsessive-compulsive disorder (OCD) patients and their core families.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed OCD patient

Exclusion Criteria:

* organic disease
* other psychiatric disorder

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: OCD patients and their parents
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-02; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Y-BOCS | Y-BOCS

CONTACTS AND LOCATIONS:
Overall Officials: Xiufeng Xu, Principal Investigator — the 1st affiliated hospital of Kunming medical college
Locations (1):
- Psychiatry department of KMC, Kunming, Yunnan, China